CLINICAL TRIAL: NCT04700553
Title: Efficacy of Localized Muscle Vibration on Lower Extremity Functional Ability in Patients With Stroke: A Randomized Controlled Trial
Brief Title: Localized Muscle Vibration Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Giuseppe Annino (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Annino, Professor, University of Rome Tor Vergata
Organization: University of Rome Tor Vergata (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 187/20
Record Dates: First submitted 2021-01-01; First posted 2021-01-08 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy intervention plus localized muscle vibration (Experimental): physical therapy intervention plus localized muscle vibration
  Interventions: Device: Localized muscle vibration; Other: Conventional physiotherapy intervention
- Conventional physical therapy intervention (Sham Comparator): physical therapy intervention
  Interventions: Other: Conventional physiotherapy intervention

INTERVENTIONS:
Device: Localized muscle vibration — All patients in both experimental and control groups received CPT protocol consisted of 30 minutes of manual resistance exercise (3 sets/10 repetitions each for knee extensors and flexors) and 30 minutes of treadmill training, short breaks (1-5 minutes) were allowed, depending on the patient tolerance. The training was conducted for 3 days per week for 8 weeks. The patients in CPT+LMV experimental group received localized muscle vibration at the end of each CPT session. The LMV was applied for 5 minutes perpendicularly along quadriceps muscle fibers. The frequency set at 30 Hz, amplitude of 2 mm.
  Other Names: manual resistance exercise; treadmill training
  Arms: Conventional physical therapy intervention plus localized muscle vibration
Other: Conventional physiotherapy intervention — All patients in both experimental and control groups received CPT protocol consisted of 30 minutes of manual resistance exercise (3 sets/10 repetitions each for knee extensors and flexors) and 30 minutes of treadmill training, short breaks (1-5 minutes) were allowed, depending on the patient tolerance. The training was conducted for 3 days per week for 8 weeks. The patients in CPT+LMV experimental group received localized muscle vibration at the end of each CPT session. The LMV was applied for 5 minutes perpendicularly along quadriceps muscle fibers. The frequency set at 30 Hz, amplitude of 2 mm.
  Other Names: manual resistance exercise; treadmill training

SUMMARY:
Background and objectives: Lower extremity functional impairments are common consequences of stroke. Thus, continuous examination of effective treatment interventions for lower extremity functions after stroke is a necessity. Localized muscle vibration (LMV) is one of the treatment interventions that incorporate sensory stimulation to improve motor cortical excitability. This study aimed to investigate the influences of 10-minutes lower extremity LMV application along with conventional physical therapy (CPT) on activities of daily living (ADL) and motor recovery on the hemiparetic lower extremity post-stroke.

Methods: A sample of 37 patients with stroke (8 females) was randomly allocated to either conventional physical therapy (CPT) control group (n=18) or conventional physical therapy and localized muscle vibration (CPT+LMV) experimental group (n=19). All patients received 3 sessions per week of CPT for 8 weeks. The CPT+LMV experimental group received 10-minute LMV at the end of each CPT session. The outcome measures used were the Barthel Index (BI), Berg Balance Scale (BBS), and goniometry for Range of Motion (ROM) assessment.

DETAILED DESCRIPTION:
All patients in both experimental and control groups received CPT protocol consisted of 30 minutes of manual resistance exercise (3 sets/10 repetitions each for knee extensors and flexors) and 30 minutes of treadmill training, short breaks (1-5 minutes) were allowed, depending on the patient tolerance. The training was conducted for 3 days per week for 8 weeks. The patients in CPT+LMV experimental group received localized muscle vibration at the end of each CPT session. The LMV was applied for 10 minutes perpendicularly along quadriceps muscle fibers. The frequency set at 30 Hz, amplitude of 2 mm.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of stroke

Exclusion Criteria:

If they had any serious orthopedic injury/disease, cardiopulmonary problems or suffered from a neurological disease (other than stroke).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Barthel Index (BI) | Change from baseline activity of daily livings at 8 weeks
  The Barthel Index of Activities of Daily Living (BI). Measure of functional disability. The BI consisting of 10 common activities of daily living (ADL) activities, administered through direct observation. These are assessed for independence/ dependence and scored via an arbitrary weighting system (originally applied to reflect nursing care and social acceptability). Eight of the ten items represent activities related to personal care; the remaining 2 are related to mobility. The index yields a total score out of 100 - the higher the score, the greater the degree of functional independence

SECONDARY OUTCOMES:
Berg Balance Scale | Change from baseline balance at 8 weeks
  The BBS provides a quantitative measure of balance. This scale consists of 14 items requiring patients to maintain their positions or complete tasks of varying levels of difficulty. All items are related to everyday life tasks. A score of zero represents an inability of the patient to complete the task and a score of 4 represents the ability of the patient to complete the task independently. The total scores range from 0 - 56. A total score of less than 45 indicates a balance impairment.
Goniometry | Change from baseline range of motion at 8 weeks
  Range of motion assessed by goniometry; is the measurement of angles, particularly those formed by joints. These angles may be measured in a standing position or in flexion or extension.
Manual Muscle Testing | Change from baseline range of motion at 8 weeks
  The MMT was used to assess muscle strength. The MMT consists of 6 grades. Grade 0 indicates no evidence of contractility (complete paralysis), and 5 indicates movement against gravity plus full resistance.
Modified Ashworth Scale | Change from baseline range of motion at 8 weeks
  The MAS was utilized to measure spasticity. The scale asses the resistance of limb to a rapid passive stretch in 6 scores from 0 to 5. Score 0 indicates normal muscle tone, and 5 indicates rigid limb.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Annino, PhD, Study Director — University of Rome Tor Vergata
Locations (1):
- Policlinico Tor Vergata, Rome, RM, Italy